CLINICAL TRIAL: NCT04839393
Title: A PHASE 1, OPEN-LABEL STUDY TO EVALUATE THE PHARMACOKINETIC INTERACTIONS BETWEEN PF-06882961 AND PF-06865571 IN HEALTHY ADULT PARTICIPANTS (PART A) AND OVERWEIGHT ADULTS OR ADULTS WITH OBESITY WHO ARE OTHERWISE HEALTHY (PART B)
Brief Title: A Drug-Drug Interaction Study Between PF-06882961 and PF-06865571 in Healthy Adult Participants and Overweight Adults or Adults With Obesity Who Are Otherwise Healthy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: C3421038
Record Dates: First submitted 2021-03-29; First posted 2021-04-09 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2022-09

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — danuglipron; ervogastat

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A - Sequence 1 (Experimental): Treatment A - PF-06882961 single dose followed by Treatment B - PF-06882961 single dose and PF-06865571 single dose
  Interventions: Drug: PF-06882961 followed by PF-06882961/PF-06865571
- Part A - Sequence 2 (Experimental): Treatment B - PF-06882961 single dose and PF-06865571 single dose followed by Treatment A - PF-06882961 single dose
  Interventions: Drug: PF-06882961/PF-06865571 followed by PF-06882961
- Part B (Experimental): Period 1: PF-06865571 single dose, Period 2: PF-06882961 twice daily dose titration, Period 3: PF-06865571 single dose and PF-06882961 twice daily dosing, Period 4: PF-06865571 twice daily dosing and PF-06882961 twice daily dosing
  Interventions: Drug: PF-06882961 + PF-06865571

INTERVENTIONS:
Drug: PF-06882961 followed by PF-06882961/PF-06865571 — Treatment A - PF-06882961 20 mg single dose followed by Treatment B - PF-06882961 20 mg single dose plus PF-06865571 300 mg single dose. There will be a washout interval between periods of at least 3 days.
  Arms: Part A - Sequence 1
Drug: PF-06882961/PF-06865571 followed by PF-06882961 — Treatment B - PF-06882961 20 mg single dose plus PF-06865571 300 mg single dose followed by Treatment A - PF-06882961 20 mg single dose. There will be a washout interval between periods of at least 3 days.
  Arms: Part A - Sequence 2
Drug: PF-06882961 + PF-06865571 — Period 1: PF-06865571 300 mg single dose (Day 1), Period 2: PF-06882961 10 mg twice daily dose titration up to 200 mg twice daily dosing (Days 3-46), Period 3: PF-06865571 300 mg single dose (Day 47) and PF-06882961 200 mg twice daily dosing (Days 47-48), Period 4: PF-06865571 300 mg twice daily dosing and PF-06882961 200 mg twice daily dosing (Days 49-62)
  Arms: Part B

SUMMARY:
This study will be conducted in 2 parts. Part A will investigate the potential effect of PF-06865571 on the pharmacokinetics (PK) of PF-06882961 in healthy adult participants. Part B will evaluate the effect of PF-06882961 on the PK of PF-06865571, as well as the effect of PF-06865571 on the PK of PF-06882961 in overweight adults or adults with obesity who are otherwise healthy.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants must be 18 to 65 years of age, inclusive, at the time of signing the ICD.

   Women can be of child-bearing potential, however, cannot be pregnant, breastfeeding, or planning to become pregnant while participating in the study.
2. Male and female participants who are overtly healthy (other than being overweight or obese in Part B only) as determined by medical evaluation including medical history, physical examination, and laboratory tests.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
4. BMI and total body weight:

   Part A: BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb); Part B: BMI ≥25 kg/m2 and not more than 40 kg/m2 at Screening; stable body weight, defined as <5 kg change (per participant report) for 90 days before Screening.
5. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy, bariatric surgery, active inflammatory bowel disease, or an intestinal resection).
3. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to COVID-19 pandemic (eg, contact with positive case, residence or travel to an area with high incidence) that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
4. Known intolerance or hypersensitivity to GLP-1 receptor agonists.
5. Known intolerance or hypersensitivity to DGAT2 inhibitors.
6. Diagnosis of type 1 or type 2 diabetes mellitus or secondary forms of diabetes at screening. Note: women with prior diagnoses of gestational diabetes during pregnancy only are eligible if they meet the other eligibility criteria.
7. History of myocardial infarction, unstable angina, arterial revascularization, stroke, New York Heart Association Functional Class II-IV heart failure, or transient ischemic attack within 6 months of Screening.
8. Any malignancy not considered cured (except basal cell carcinoma and squamous cell carcinoma of the skin); a study participant is considered cured if there has been no evidence of cancer recurrence in the previous 5 years (from Screening).
9. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2, or study participants with suspected medullary thyroid carcinoma per the investigator's judgment.
10. Acute pancreatitis or history of chronic pancreatitis.
11. Symptomatic gallbladder disease.
12. Medical history or characteristics suggestive of genetic or syndromic obesity or obesity induced by other endocrinological disorders (eg, Cushing Syndrome).
13. History of major depressive disorder or history of other severe psychiatric disorders (eg, schizophrenia or bipolar disorder) within the last 2 years from screening.
14. Known medical history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic active hepatitis B or C, primary biliary cirrhosis, alcoholic liver disease, primary sclerosing cholangitis, autoimmune hepatitis, overlap syndrome, or prior known drug-induced liver injury.
15. History of HIV infection.
16. Any lifetime history of a suicide attempt.
17. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
18. Prohibited prior/concomitant medication as per protocol.
19. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer). An emergency use authorized or approved COVID-19 vaccine is considered a concomitant medication.
20. Known prior participation in a clinical trial with PF-06882961 or PF-06865571.
21. Part B only: A Patient Health Questionnaire (PHQ-9) score ≥15 obtained at Screening or Day -1.
22. Part B only: Response of "yes" to question 4 or 5, or on any behavioral question on the C-SSRS at Screening or Day -1.
23. A positive urine drug test.
24. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
25. Screening 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTc interval >450 msec, complete LBBB, signs of an acute or indeterminate-age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third-degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate-corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
26. A positive COVID-19 test at or after screening.
27. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary: HbA1c ≥6.5%. AST or ALT > ULN. Total bilirubin level > ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and are eligible for this study provided the direct bilirubin level is ≤ ULN.

    TSH > ULN or < LLN. Serum calcitonin > ULN. Amylase or lipase > ULN. Fasting blood glucose ≥126 mg/dL. Fasting triglycerides >200 mg/dL. INR > ULN. PLT < LLN. eGFR <80 mL/min/1.73 m2 as calculated by the CKD-EPI equation. Positive testing for HIV, HepBsAg, or HCVAb. Study participants positive for HCVAb are to be excluded unless known to have been treated with a known curative therapy and negative for HCV RNA. Hepatitis B vaccination is allowed.
28. Participation in a formal weight reduction program (eg, Weight Watchers) within 90 days prior to Screening.
29. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
30. Current use of tobacco or nicotine containing products in excess of the equivalent of 5 cigarettes per day.
31. Known or suspected illicit drug use.
32. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dose randomization (Day -1).
33. History of sensitivity to heparin or heparin-induced thrombocytopenia if Hep-lock is used for IV blood draw.
34. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
35. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Orange County Research Center, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3421038

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 participants were enrolled in Part A of the study and 19 participants were enrolled in Part B of the study.
Pre-assignment Details: Part A of the study was an open-label, 2-period, 2-sequence, crossover study. Part B of the study was an open-label, fixed-sequence study.
Groups:
- Part A Sequence 1: There were 2 periods in Part A. Participants assigned to Sequence 1 received a single dose of PF-06882961 20 mg in Period 1, after a washout of at least 3 days, participants received a single dose of PF-06882961 20 mg + PF-06865571 300 mg in Period 2.
- Part A Sequence 2: There were 2 periods in Part A. Participants assigned to Sequence 2 received a single dose of PF-06882961 20 mg + PF-06865571 300 mg in Period 1, after a washout of at least 3 days, participants received a single dose of PF-06882961 20 mg in Period 2.
- Part B: There were 4 periods in Part B. All participants in Part B received a single dose of PF-06865571 300 mg on Day 1 Period 1 (Days 1-2) , and PF-06882961 10 mg twice daily (BID) titrated to 200 mg BID in Period 2 (Days 3-46). In Period 3 (Days 47-48), participants received a single dose of PF-06865571 300 mg on Day 47 only and PF-06882961 200 mg BID. In Period 4 (Days 49-62), participants received PF-06865571 300 mg BID and PF-06882961 200 mg BID on Days 49-61.
Period: Overall Study
Arm/Group | Part A Sequence 1 | Part A Sequence 2 | Part B
Started | 4 | 4 | 19
Received Treatment | 4 | 4 | 19
Completed | 4 | 4 | 16
Not Completed | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Withdrawal by participant | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A Sequence 1 | Part A Sequence 2 | Part B | Total
Number analyzed (Participants) | 4 | 4 | 19 | 27
Age, Customized [Number; unit: Participants]
  18-44 Years | 3 | 3 | 7 | 13
  45-64 Years | 1 | 1 | 12 | 14
  >=65 Years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 3 | 3 | 18 | 24
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 2 | 1 | 15 | 18
  Black or African American | 2 | 3 | 4 | 9
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 1 | 1 | 5 | 7
  Not Hispanic or Latino | 3 | 3 | 14 | 20

OUTCOME MEASURES:

1. Primary Outcome: Part A: PF-06882961 Maximum Observed Concentration (Cmax)
Description: Cmax for PF-06882961 was observed directly from data.
Time Frame: 0 (prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16 and 24 hours post-dose on Day 1
Population: The PK concentration analysis set for PF-06882961 included all randomized participants who received at least 1 dose of PF-06882961 and in whom at least 1 plasma concentration value was reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- PF-06882961 20 mg: Participants received PF-06882961 20 mg on Day 1 in either Period 1 or 2, depending on the treatment sequence they were assigned to.
- PF-06882961 20 mg + PF-06865571 300 mg: Participants received PF-06882961 20 mg + PF-06865571 300 mg on Day 1 in either Period 1 or 2, depending on the treatment sequence they were assigned to.
Arm/Group | PF-06882961 20 mg | PF-06882961 20 mg + PF-06865571 300 mg
Number analyzed (Participants) | 8 | 8
nanogram per milliliter (ng/mL) | 15.69 (198) | 17.09 (265)
Statistical Analysis 1: Comparison: PF-06882961 20 mg vs PF-06882961 20 mg + PF-06865571 300 mg; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; Mixed Models Analysis; Adjusted Geometric Mean Ratio (%) = 108.86, 90% CI 2-sided [87.24 to 135.84]

2. Primary Outcome: Part A: PF-06882961 Area Under the Plasma Concentration-time Profile From Time 0 to the Time 24 Hours Post-dose (AUC24)
Description: AUC24 for PF-06882961 was determined by Linear/Log trapezoidal method.
Time Frame: 0 (prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16 and 24 hours post-dose on Day 1
Population: The PK parameter analysis set for PF-06882961 included all randomized participants who received at least 1 dose of PF-06882961 and in whom at least 1 parameter value was reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng.hr/mL)
Groups:
- PF-06892961 20 mg + PF-06865571 300 mg: Participants received PF-06882961 20 mg + PF-06865571 300 mg on Day 1 in either Period 1 or 2, depending on the treatment sequence they were assigned to.
Arm/Group | PF-06882961 20 mg | PF-06892961 20 mg + PF-06865571 300 mg
Number analyzed (Participants) | 8 | 8
nanogram*hour per milliliter (ng.hr/mL) | 109.5 (198) | 123.9 (311)
Statistical Analysis 1: Comparison: PF-06882961 20 mg vs PF-06892961 20 mg + PF-06865571 300 mg; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; Mixed Models Analysis; Adjusted Geometric Mean Ratio = 113.14, 90% CI 2-sided [89.34 to 143.28]

3. Primary Outcome: Part B: PF-06865571 Cmax on Day 1 and Day 47
Description: Cmax for PF-06865571 was observed directly from data on Day 1 and Day 47.
Time Frame: 0 (prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 24 and 48 hours post-dose
Population: The PK concentration analysis set for PF-06865571 included all randomized participants who received at least 1 dose of PF-06865571 and in whom at least 1 plasma concentration value is reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Day 1 (PF-06865571 300 mg); Day 47 (PF-06865571 300 mg + PF-06882961 200 mg BID): All participants in Part B received a single dose of PF-06865571 300 mg on Day 1 Period 1 (Days 1-2) , and PF-06882961 10 mg twice daily (BID) titrated to 200 mg BID in Period 2 (Days 3-46). In Period 3 (Days 47-48), participants received a single dose of PF-06865571 300 mg on Day 47 only and PF-06882961 200 mg BID. In Period 4, participants received PF-06865571 300 mg BID and PF-06882961 200 mg BID on Days 49-61.
Arm/Group | Day 1 (PF-06865571 300 mg) | Day 47 (PF-06865571 300 mg + PF-06882961 200 mg BID)
Number analyzed (Participants) | 19 | 16
ng/mL | 2078 (37) | 791 (41)
Statistical Analysis 1: Comparison: Day 1 (PF-06865571 300 mg) vs Day 47 (PF-06865571 300 mg + PF-06882961 200 mg BID); The test treatment was PF-06865571 300 mg + PF-06882961 200 mg BID (Period 3 - Day 47), which was reported separately in comparison to the reference treatment of PF-06865571 300 mg (Period 1 - Day 1); Test type: Other — The ratio and 90% confidence interval were expressed as percentages; Mixed Models Analysis; Adjusted Geometric Mean Ratio = 38.73, 90% CI 2-sided [32.80 to 45.74]

4. Primary Outcome: Part B: PF-06865571 Area Under the Plasma Concentration-time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) on Day 1 and Day 47
Description: AUClast for PF-06865571 was determined by Linear/Log trapezoidal method on Day 1 and Day 47.
Time Frame: 0 (prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 24 and 48 hours post-dose
Population: The PK parameter analysis set for PF-06865571 included all randomized participants who received at least 1 dose of PF-06865571 and in whom at least 1 parameter value was reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Day 1 (PF-06865571 300 mg) | Day 47 (PF-06865571 300 mg + PF-06882961 200 mg BID)
Number analyzed (Participants) | 19 | 16
ng*hr/mL | 9011 (38) | 6630 (40)
Statistical Analysis 1: Comparison: Day 1 (PF-06865571 300 mg) vs Day 47 (PF-06865571 300 mg + PF-06882961 200 mg BID); Test type: Other — The ratio and 90% confidence interval were expressed as percentages; Mixed Models Analysis; Adjusted Geometric Mean Ratio = 73.91, 90% CI 2-sided [67.95 to 80.40]

5. Primary Outcome: Part B: PF-06865571 Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) on Day 1 and Day 47
Description: AUCinf for PF-06865571 was calculated as AUClast + (Clast*/kel) on Day 1 and Day 47. Clast* was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis and kel was the elimination rate constant.
Time Frame: 0 (prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 24 and 48 hours post-dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Day 1 (PF-06865571 300 mg) | Day 47 (PF-06865571 300 mg + PF-06882961 200 mg BID)
Number analyzed (Participants) | 19 | 14
ng*hr/mL | 9029 (38) | 6726 (43)
Statistical Analysis 1: Comparison: Day 1 (PF-06865571 300 mg) vs Day 47 (PF-06865571 300 mg + PF-06882961 200 mg BID); Test type: Other — The ratio and 90% confidence interval were expressed as percentages; Mixed Models Analysis; Adjusted Geometric Mean Ratio = 73.20, 90% CI 2-sided [66.82 to 80.18]

6. Primary Outcome: Part B: PF-06882961 Cmax on Day 46 and Day 61
Description: Cmax for PF-06882961 was observed directly from data on Day 46 and Day 61.
Time Frame: 0 (prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Day 46 (PF-06882961 Titration up to 200 mg BID); Day 61 (PF-06865571 300 mg BID + PF-06882961 200 mg BID): All participants in Part B received a single dose of PF-06865571 300 mg on Day 1 Period 1 (Days 1-2) , and PF-06882961 10 mg twice daily (BID) titrated to 200 mg BID in Period 2 (Days 3-46). In Period 3 (Days 47-48), participants received a single dose of PF-06865571 300 mg on Day 47 only and PF-06882961 200 mg BID. In Period 4, participants received PF-06865571 300 mg BID and PF-06882961 200 mg BID on Days 49-61.
Arm/Group | Day 46 (PF-06882961 Titration up to 200 mg BID) | Day 61 (PF-06865571 300 mg BID + PF-06882961 200 mg BID)
Number analyzed (Participants) | 15 | 14
ng/mL | 1187 (115) | 1393 (107)
Statistical Analysis 1: Comparison: Day 46 (PF-06882961 Titration up to 200 mg BID) vs Day 61 (PF-06865571 300 mg BID + PF-06882961 200 mg BID); Test type: Other — The ratio and 90% confidence interval were expressed as percentages; Mixed Models Analysis; Adjusted Geometric Mean Ratio = 115.30, 90% CI 2-sided [85.37 to 155.73]

7. Primary Outcome: Part B: PF-06882961 Area Under the Plasma Concentration-time Profile From Time 0 to the Time 12 Hours Post-dose (AUC12) on Day 46 and Day 61
Description: AUC 12 for PF-06882961 was determined by Linear/Log trapezoidal method on Day 46 and Day 61.
Time Frame: 0 (prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hr/mL
Arm/Group | Day 46 (PF-06882961 Titration up to 200 mg BID) | Day 61 (PF-06865571 300 mg BID + PF-06882961 200 mg BID)
Number analyzed (Participants) | 15 | 14
ng.hr/mL | 7682 (99) | 9312 (99)
Statistical Analysis 1: Comparison: Day 46 (PF-06882961 Titration up to 200 mg BID) vs Day 61 (PF-06865571 300 mg BID + PF-06882961 200 mg BID); Test type: Other — The ratio and 90% confidence interval were expressed as percentages; Mixed Models Analysis; Adjusted Geometric Mean Ratio = 118.64, 90% CI 2-sided [94.05 to 149.66]

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) in Part A
Description: An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Any AEs occurring following start of study intervention were counted as treatment emergent. Serious AEs (SAEs) were defined as any untoward medical occurrence at any dose that resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or caused prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduction normal life functions). AEs included SAEs and non-serious AEs. Relatedness to study treatment was determined by the investigator.
Time Frame: Up to 68 days
Population: The safety analysis set included all participants randomly assigned to investigational product and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06882961 20 mg | PF-06882961 20 mg + PF-06865571 300 mg
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities in Part A
Description: Safety laboratory assessments included clinical chemistry, hematology, urinalysis, and other tests. Abnormality was determined at the investigator's discretion. Abnormalities without regard to baseline abnormalities were reported.
Time Frame: From Screening (28 days prior to the day of treatment) to Day 2 of Period 2, for a maximum of 33 Days
Population: The safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable laboratory values were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06882961 20 mg | PF-06882961 20 mg + PF-06865571 300 mg
Number analyzed (Participants) | 8 | 8
Participants | 2 | 3

10. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Pre-specified Criteria in Part A
Description: Single, supine vital signs assessments included systolic blood pressure (BP), diastolic BP and pulse rate. Abnormality in vital signs included: pulse rate <40 beats per minute (bpm) or >120bpm; supine diastolic BP <50 millimeter of mercury (mmHg), increase and decrease in change from baseline (BL) of >=20mmHg; supine systolic blood pressure <90mmHg, increase and decrease in change from BL of >=30mmHg.
Time Frame: From Screening (28 days prior to the day of treatment) to Day 2 of Period 2, for a maximum of 33 Days
Population: The safety analysis set included all participants randomly assigned to investigational product and who took at least 1 dose of study intervention. Participants with evaluable vital signs data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06882961 20 mg | PF-06882961 20 mg + PF-06865571 300 mg
Number analyzed (Participants) | 8 | 8
Participants
  Supine systolic BP value <90mmHg | 0 | 0
  Supine systolic BP change >=30mmHg increase | 0 | 0
  Supine systolic BP change >=30mmHg decrease | 0 | 1
  Supine diastolic BP value <50mmHg | 0 | 0
  Supine diastolic BP change >=20mmHg increase | 0 | 0
  Supine diastolic BP change >=20mmHg decrease | 0 | 0
  Pulse rate value <40bpm | 0 | 0
  Pulse rate value >120bpm | 0 | 0

11. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Pre-specified Criteria in Part A
Description: ECG assessments included pulse rate (PR), QT, QTcF intervals and QRS complex. ECG abnormalities criteria included: PR interval value >= 300msec, or baseline (BL) >200msec and >=25% increase from BL, or BL <=200msec and >=50% increase from BL; QRS interval value >= 140msec, or percent change from BL >=50%; QTcF value >400 and <=480msec, or >480 and <=500 msec, or >500msec, or change from BL>30 and <=60msec, or change from BL >60msec.
Time Frame: From Screening (28 days prior to the day of treatment) to Day 2 of Period 2, for a maximum of 33 Days
Population: The analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable ECG data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06882961 20 mg | PF-06882961 20 mg + PF-06865571 300 mg
Number analyzed (Participants) | 8 | 8
Participants
  PR interval value >= 300 msec | 0 | 0
  PR interval %change >=25/50% (BL >200 msec and >=25% increase or BL <=200 msec and >=50% increase) | 0 | 0
  QRS interval value>=140 msec | 0 | 0
  QRS interval %change >=50% | 0 | 0
  QTcF value >450 and <=480 msec | 0 | 0
  QTcF value >480 and <=500 msec | 0 | 0
  QTcF value >500 msec | 0 | 0
  QTcF change >30 and <=60 msec | 0 | 0
  QTcF change >60 msec | 0 | 0

12. Secondary Outcome: Number of Participants With TEAEs in Part B
Description: as for outcome 8
Time Frame: Up to 173 days
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- PF-06865571 300 mg; PF-06882961 Titration up to 200 mg BID; PF-06865571 300 mg + PF-06882961 200 mg BID; PF-06865571 300 mg BID + PF-06882961 200 mg BID: All participants in Part B received a single dose of PF-06865571 300 mg on Day 1 Period 1 (Days 1-2) , and PF-06882961 10 mg twice daily (BID) titrated to 200 mg BID in Period 2 (Days 3-46). In Period 3 (Days 47-48), participants received a single dose of PF-06865571 300 mg on Day 47 only and PF-06882961 200 mg BID. In Period 4, participants received PF-06865571 300 mg BID and PF-06882961 200 mg BID on Days 49-61.
Arm/Group | PF-06865571 300 mg | PF-06882961 Titration up to 200 mg BID | PF-06865571 300 mg + PF-06882961 200 mg BID | PF-06865571 300 mg BID + PF-06882961 200 mg BID
Number analyzed (Participants) | 19 | 19 | 16 | 16
Participants
  All-causality TEAEs | 1 | 18 | 6 | 10
  Treatment-related TEAEs | 1 | 16 | 6 | 10

13. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities in Part B
Description: as for outcome 9
Time Frame: From Screening (28 days prior to follow-up visit (up to 10 days after the last dose of treatment), for a maximum of 148 Days
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06865571 300 mg | PF-06882961 Titration up to 200 mg BID | PF-06865571 300 mg + PF-06882961 200 mg BID | PF-06865571 300 mg BID + PF-06882961 200 mg BID
Number analyzed (Participants) | 19 | 19 | 16 | 16
Participants | 0 | 16 | 0 | 15

14. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Pre-specified Criteria in Part B
Description: Single, supine vital signs assessments included systolic blood pressure (BP), diastolic BP and pulse rate. Abnormality in vital signs included: pulse rate <40 beats per minute (bpm) or >120bpm; supine diastolic BP <50 millimeter of mercury (mmHg), increase and decrease in change from BL of >=20mmHg; supine systolic blood pressure <90mmHg, increase and decrease in change from BL of >=30mmHg.
Time Frame: as for outcome 13
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06865571 300 mg | PF-06882961 Titration up to 200 mg BID | PF-06865571 300 mg + PF-06882961 200 mg BID | PF-06865571 300 mg BID + PF-06882961 200 mg BID
Number analyzed (Participants) | 19 | 19 | 16 | 16
Participants
  Supine systolic BP value <90mmHg | 0 | 0 | 0 | 0
  Supine systolic BP change >=30mmHg increase | 0 | 0 | 0 | 0
  Supine systolic BP change >=30mmHg decrease | 0 | 0 | 0 | 0
  Supine diastolic BP value <50mmHg | 0 | 0 | 0 | 0
  Supine diastolic BP change >=20mmHg increase | 0 | 1 | 0 | 1
  Supine diastolic BP change >=20mmHg decrease | 0 | 0 | 0 | 0
  Pulse rate value <40bpm | 0 | 0 | 0 | 0
  Pulse rate value >120bpm | 0 | 0 | 0 | 0

15. Secondary Outcome: Change From Baseline in Body Weight for Participants in Part B
Description: Changes from baseline in body weight of the participants were measured.
Time Frame: At Baseline (Days -28 to 2), on Period 2, Days 6, 13, 20 ,27, 34, and 41, Period 4, Days 9 and14 and follow-up visit (Days 68-71)
Population: The analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable body weight data were analyzed.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Groups:
- All Participants: All participants in Part B received a single dose of PF-06865571 300 mg on Day 1 Period 1 (Days 1-2) , and PF-06882961 10 mg twice daily (BID) titrated to 200 mg BID in Period 2 (Days 3-46). In Period 3 (Days 47-48), participants received a single dose of PF-06865571 300 mg on Day 47 only and PF-06882961 200 mg BID. In Period 4, participants received PF-06865571 300 mg BID and PF-06882961 200 mg BID on Days 49-61.
Arm/Group | All Participants
Number analyzed (Participants) | 19
kilogram (kg)
  Period 2 Day 6 | -0.73 (1.999)
  Period 2 Day 13 | -1.49 (2.260)
  Period 2 Day 20 | -2.48 (2.242)
  Period 2 Day 27 | -3.32 (2.525)
  Period 2 Day 34 | -4.76 (3.141)
  Period 2 Day 41 | -5.39 (2.599)
  Period 4 Day 2 | -6.09 (3.088)
  Period 4 Day 9 | -6.89 (3.299)
  Period 4 Day 14 | -6.93 (3.632)
  Follow-up | -4.59 (3.916)

16. Secondary Outcome: Number of Participants With ECG Data Meeting Pre-specified Criteria in Part B
Description: ECG assessments included PR, QT, QTcF intervals and QRS complex. ECG abnormalities criteria included: PR interval value >= 300msec, or BL >200msec and >=25% increase from BL, or BL <=200msec and >=50% increase from BL; QRS interval value >= 140msec, or percent change from BL >=50%; QTcF value >400 and <=480msec, or >480 and <=500 msec, or >500msec, or change from BL>30 and <=60msec, or change from BL >60msec.
Time Frame: as for outcome 13
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06882961 Titration up to 200 mg BID | PF-06865571 300 mg BID + PF-06882961 200 mg BID
Number analyzed (Participants) | 19 | 16
Participants
  PR interval value>=300 msec | 0 | 1
  PR interval %change >=25/50% (BL >200 msec and >=25% increase or BL <=200 msec and >=50% increase) | 0 | 0
  QRS interval value>=140 msec | 0 | 0
  QRS interval %change >=50% | 0 | 0
  QTcF value >450 and <=480 msec | 0 | 0
  QTcF value >480 and <=500 msec | 0 | 0
  QTcF value >500 msec | 0 | 0
  QTcF change >30 and <=60 msec | 0 | 0
  QTcF change >60 msec | 0 | 0

17. Secondary Outcome: Number of Participants With Suicidal Ideation or Behavior as Per C-SSRS Mapped to Columbia Classification Algorithm of Suicide Assessment (C-CASA) in Part B
Description: The C-SSRS was an interview-based rating scale to systematically assess suicidal ideation and suicidal behavior. C-SSRS assessed whether participant experienced any of the following 1: completed suicide, 2: suicide attempt (response of "yes" on "actual attempt"), 3: preparatory acts toward imminent suicidal behavior ("yes" on "aborted attempt", "interrupted attempt", "preparatory acts or behavior"), 4: any suicidal behavior or ideation, suicidal ideation ("yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent"), 7: self-injurious behavior, no suicidal intent ("yes" on "has participant engaged in non-suicidal self-injurious behavior").
Time Frame: At Screening (Days -28 to -2), Baseline (Period 1 Day -1), on Period 2, Days 6, 13, 20, 27, 34 and 41, Period 4, Days 2, 9 and 14 and follow-up visit (Days 68-71)
Population: The analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable C-SSRS results were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 19
Participants
  Baseline | 0
  Period 2 Day 6 | 0
  Period 2 Day 13 | 0
  Period 2 Day 20 | 0
  Period 2 Day 27 | 0
  Period 2 Day 34: number analyzed (Participants) | 16
  Period 2 Day 34 | 0
  Period 2 Day 41: number analyzed (Participants) | 16
  Period 2 Day 41 | 0
  Period 4 Day 2: number analyzed (Participants) | 16
  Period 4 Day 2 | 0
  Period 4 Day 9: number analyzed (Participants) | 16
  Period 4 Day 9 | 0
  Period 4 Day 14: number analyzed (Participants) | 16
  Period 4 Day 14 | 0
  Follow-up: number analyzed (Participants) | 16
  Follow-up | 0

18. Secondary Outcome: Number of Participants With Response to PHQ-9 in Part B
Description: The PHQ-9 is a 9 item self-report scale for the assessment of depressive symptoms. The questions included "little interest/pleasure in things", "feeling down depressed or hopeless", "trouble falling or staying asleep", "feeling tired or little energy", "poor appetite or overeating", "feeling bad about yourself", "trouble concentrating on things", "moving slowly or fidgety/restless" and "thoughts you be better off dead". Each item was scored on scale of "not at all", "several days", "more than half the days" to "nearly every day". Total score range: 0-27 (each item with scale from 0 [not at all] to 3 [nearly every day]. Higher score=greater severity). Any participant with a response of any scale other than "not at all" to any of the 9 questions was counted.
Time Frame: as for outcome 17
Population: The analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable PHQ-9 results were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 19
Participants
  Baseline | 2
  Period 2 Day 6 | 0
  Period 2 Day 13 | 0
  Period 2 Day 20 | 0
  Period 2 Day 27 | 0
  Period 2 Day 34: number analyzed (Participants) | 16
  Period 2 Day 34 | 0
  Period 2 Day 41: number analyzed (Participants) | 16
  Period 2 Day 41 | 0
  Period 4 Day 2: number analyzed (Participants) | 16
  Period 4 Day 2 | 0
  Period 4 Day 9: number analyzed (Participants) | 16
  Period 4 Day 9 | 0
  Period 4 Day 14: number analyzed (Participants) | 16
  Period 4 Day 14 | 0
  Follow-up: number analyzed (Participants) | 16
  Follow-up | 0

ADVERSE EVENTS:
Time Frame: Up to 68 days for Part A and up to 173 days for Part B.
Groups:
- PF-06882961 20 mg + PF-06865571 300 mg: In Part A, participants received PF-06882961 20 mg + PF-06865571 300 mg on Day 1 in either Period 1 or 2, depending on the treatment sequence they were assigned to.
- PF-06865571 300 mg: Participants received a single dose of PF-06865571 300 mg on Day 1 in Part B Period 1 (Days 1-2).
- PF-06882961 Titration up to 200 mg BID: Participants received PF-06882961 titrated up to 200 mg BID in Part B Period 2 (Days 3-46).
- PF-06865571 300 mg + PF-06882961 200 mg BID: Participants received PF-06865571 300 mg single dose on Day 47 and PF-06882961 200 mg BID in Period 3 (Days 47-48).
- PF-06865571 300 mg BID + PF-06882961 200 mg BID: Participants received PF-06865571 300 mg BID and PF-06882961 200 mg BID in on Days 49-61 in Period 4.
Arm/Group | PF-06882961 20 mg | PF-06882961 20 mg + PF-06865571 300 mg | PF-06865571 300 mg | PF-06882961 Titration up to 200 mg BID | PF-06865571 300 mg + PF-06882961 200 mg BID | PF-06865571 300 mg BID + PF-06882961 200 mg BID
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/19 | 0/19 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/19 | 0/19 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 1/19 | 18/19 | 6/16 | 10/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06882961 20 mg (N=8) | PF-06882961 20 mg + PF-06865571 300 mg (N=8) | PF-06865571 300 mg (N=19) | PF-06882961 Titration up to 200 mg BID (N=19) | PF-06865571 300 mg + PF-06882961 200 mg BID (N=16) | PF-06865571 300 mg BID + PF-06882961 200 mg BID (N=16)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 6 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 8 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 12 | 1 | 6
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 7 | 3 | 6
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 3 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 10 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 4 | 1 | 4
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 8 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT04839393/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT04839393/SAP_001.pdf